CLINICAL TRIAL: NCT05355493
Title: The Effect of Mental Fatigue on the Cerebral Oxygenation During Endurance Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Jonas De Wachter, Principal Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: NIRS_EX
Record Dates: First submitted 2022-02-08; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Mental Fatigue; Near Infrared Spectroscopy; NIRS; Condition; Cerebral Heamodynamics
Keywords: NIRS; Time to exhaustion; Prefrontal cortex; Cerebral oxygenation
MeSH Terms: conditions — Mental Fatigue; Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Mental Fatigue condition (Experimental): A Stroop task, of approximately 60 min, partitioned in 6 blocks of 336 stimuli, will be used as the mentally fatiguing task. In this task, four colored words ("rood", "blauw", "groen" and "geel") will be presented one at a time on a computer screen. The participants will be required to indicate the color of the word, ignoring the meaning of the word itself. If, however, the ink color is red, the button to be pressed will be the button linked to the real meaning of the word, not the ink color. The word presented and its ink color will be randomly selected by the computer (100% incongruent), with all incongruent word-color combinations being equally common (meaning, in each block 84 words will be presented in the color red, yellow, green and blue). Subjects will be instructed to respond as quickly and accurately as possible. To assess performance accuracy (ACC) and reaction time (RT) will be collected and averaged every block.
  Interventions: Behavioral: Time to Exhaustion cycling test; Behavioral: Go/NoGo task
- Control condition (Active Comparator): In the control task subjects will have to watch a documentary during 60 min on the same computer screen as that used for the experimental trial. In order to avoid under- and over-arousal the subjects will have the opportunity to choose between several episodes (One Planet, Frozen Worlds, Jungles, Costal Seas, From Desserts to Grasslands, The High Seas, Fresh Water and Forests) of the Netflix documentary "Our Planet, 2019" as proposed by the research team. During the control task physiological and psychological measures will be assessed at the same time points as during the mental fatigue trial.
  Interventions: Behavioral: Time to Exhaustion cycling test; Behavioral: Go/NoGo task

INTERVENTIONS:
Behavioral: Time to Exhaustion cycling test — After completing the MF/control task. Participants will be asked to take place on the cycle ergometer. Participants will perform a 3-min warm-up at 40% of peak power output followed by a rectangular workload at a power output corresponding to their predetermined respiratory compensation point (±80% PPO). RPM was freely chosen between 60 and 100 RPM and was recorded every minute. TTE was measured from the start until the pedal frequency was less than 60 RPM for more than 5s. This TTE task was chosen, based on a previous study of Marcora et al. (2009), who found that mental fatigue impairs physical performance. A researcher will sit behind the subject to ensure compliance with treatment. Subjects will be equipped with a heart rate monitor to continuously follow up heart rate. Subjective psychological assessment will take place with a M-VAS-scale, the NASA-TLX, the success motivation and intrinsic motivation scales, Karolinska Sleepiness Scale and visual analog scale for boredom.
Behavioral: Go/NoGo task — Participants are to react to different stimuli displayed on a computer screen, preceded by a screen with general instructions. Two different stimuli were present at the same time: a Go or NoGo stimulus, and a left or right stimulus (meaning that four combinations are possible: GoRight, GoLeft, NoGoRight and NoGoLeft). If a Go-stimulus is presented, participants are instructed to react to the left or right stimuli with the corresponding arrows. However, if a NoGo stimulus is presented, participants are instructed to refrain from reacting to the either the left or right stimuli. This proposed paradigm measures attention, response inhibition and working memory. Stimuli will be presented for 500 ms, with a varying interstimulus time between 1100 and 1700 ms. Outcomes for Go trials include reaction time and accuracy while the outcome for NoGo trials is only accuracy.

SUMMARY:
The experiment will consist of 3 consecutive trials performed in a sound-insulated climate chamber (20°C and 40% RH) at the VUB. Participants will be asked to return 3 successive weeks. Trained staff (pre-doctoral researchers and trained master students) will be present during the experimental trials. The first visit will be a familiarization trial in which they will complete all procedures as if it was an experimental trial, except for the interventional 60min Stroop task. Instead of the 60-min Stroop task the participants' maximal cognitive capacity will be determined.

The participant wil come in, perform a cognitive performance test, will then perform the intervention/control procedure, which will be followed by an additional conduction of the same cognitive performance test as before the intervention/control, as well as a physical performance test (time to exhaustion cycling test). The intervention will consist of a 60 min Stroop task, while the control trial will consist of watching a documentary of the same duration. Multiple different questionnaires (e.g. to assess the mentally fatigued state of participants) will be assessed throughout the experimental/control trial. The aim of this study will be to research if mental fatigue influences prefrontal cortex oxygenation during a time to exhaustion cycling test. Marcora et al. (2009) already showed a decrease in cycling performance during the exact same protocol.

DETAILED DESCRIPTION:
The investigators use a randomized, blinded, placebo controlled, counter-balanced, cross-over design. The real purpose of the study will be hold back from the participants by recruiting participants who are unaware of the possible negative effects of mental fatigue. We will inform the participants in a way that explains the study as an investigation about the influence of different cognitive tasks on a subsequent cycling. the investigators will strive equal expectations for all the participants in both the experimental and the control trial concerning the influence of the cognitive task on the cognitive and cycling task. At the end of the last trial the investigators will ask a standardized question to follow up on their thoughts about the objective of the study.

The experiment will consist of 3 consecutive trials performed in a sound-insulated climate chamber (20°C and 40% RH) at the VUB. Participants will be asked to return 3 successive weeks. Trained staff (pre-doctoral researchers and trained master students) will be present during the experimental trials. During the first visit, subjects will read and sign the informed consent and get a thorough explanation of what is expected from them, afterwards they will have the possibility to ask questions. After signing, participants complete a familiarization trial in which they will complete all procedures as if it was an experimental trial, except for the 60min cognitive task. Instead of the 60-min cognitive task the participants' maximal cognitive capacity will be determined. Therefore, a Stroop task divided in blocks of 96 stimuli will be used. After each block, the accuracy (ACC) will be calculated. When the ACC is higher than 85%, the difficulty of the Stroop task will be increased by decreasing the stimulus presentation time (SPT). If the ACC is lower than 85%, this block will be considered as an 'error' and the subject must re-do the block without changing the SPT. The first block will have a SPT of 1500 ms and will have the main objective to get familiar with the task. When the required accuracy is achieved, the SPT will decrease in the following order: 1100, 900, 800, 700, 650, 600, 550 ms… to determine the individual cognitive load. Before the start of each block, the subjects will be able to take a break if they like. When the subject makes three errors in a row, or five errors during the whole trial, the trial is considered as completed and will be ended. The SPT of the last, successfully completed block will be considered as the maximum capacity of that individual and will be used to individualize the difficulty of the 60-min Stroop task. There will be a continuous feedback of the performance to motivate the subjects, as this has been pointed out by Kurzban et al. to be important for task-engagement.

The next two trials will be performed in a counterbalanced randomized order, a mental fatigue trial (MF) and a control trial (CON). Randomization will be assured by using a web-based computer program (www.randomization.com) to determine treatment order (MF or CON trial; see intervention for details). All trials will be separated by at least 5 days to ensure full recovery.

After arrival at the laboratory for the experimental trials, participants will be asked to go to the toilet, after which they enter the climatic chamber which has reached 20°C and 40%RH. Participants will have to fill in 2 questionnaires (~3min) to estimate mood and motivation. NIRS equipment will be applied. The NIRS-optode pair will be applied prefrontally. NIRS measurement will start to verify hemodynamic changes during the absorption period. Physiological measures (HR, SaO2, BP, Hb, Respiratory Rate (RR), Glucose, NIRS, ventilation (VE), Blood lactate (BL) will be recorded.

Go/NoGo. As a manipulation check, the Go/NoGo paradigm task will be used to assess cognitive performance as suggested by Guo et al. (2018) and Kato et al. (2009). Participants are to react to different stimuli displayed on a computer screen positioned about 1 meter from the subject, preceded by a screen with general instructions. Two different stimuli were present at the same time: a Go or NoGo stimulus, and a left or right stimulus (meaning that four combinations are possible: GoRight, GoLeft, NoGoRight and NoGoLeft). If a Go-stimulus is presented, participants are instructed to react to the left or right stimuli with the corresponding arrows. However, if a NoGo stimulus is presented, participants are instructed to refrain from reacting to the either the left or right stimuli. This proposed paradigm measures attention, response inhibition and working memory, executive functions who are all consistently negatively impacted by MF. Stimuli will be presented for 500 ms, with a varying interstimulus time between 1100 and 1700 ms. Outcomes for Go trials include reaction time and accuracy while the outcome for NoGo trials is only accuracy. The ratio of Go/NoGo trials will be 80 to 20% respectively. Since the trials concern seven different interstimulus times, 1 cycle of trials consists of 56 Go and 14 NoGo trials. Moreover, to consistently detect large ERP's, research has suggested that between 30 and 40 stimuli should be present. Therefore, to be able to investigate ERP's in NoGo trials, at least 3 cycles are necessary to complete, leading to a tot task duration of about 6,5 min (taken into account a mean trial duration of 1900 ms).

Mental fatigue task:

A modified Stroop task, based on their performance during max test (familiarization session) of approximately 60 min, partitioned in 6 blocks of 336 stimuli, will be used as the mentally fatiguing task. In this task, four colored words ("rood", "blauw", "groen" and "geel") will be presented one at a time on a computer screen. The participants will be required to indicate the color of the word, ignoring the meaning of the word itself. If, however, the ink color is red, the button to be pressed will be the button linked to the real meaning of the word, not the ink color. The word presented and its ink color will be randomly selected by the computer (100% incongruent), with all incongruent word-color combinations being equally common (meaning, in each block 84 words will be presented in the color red, yellow, green and blue). Each word will be presented on screen in 34 point font for 1000 ms with an inter-stimulus interval based on their performance on the max test. Subjects will be instructed to respond as quickly and accurately as possible. To assess performance accuracy (ACC) and reaction time (RT) will be collected and averaged every block. Each of the 6 blocks will be separated by a 30-s period during which stimuli will keep presenting themselves, but where the researchers will assess the mental fatigue visual analog scale (M-VAS). Subjects will be asked to draw a line with their dominant hand on the M-VAS and to continue answering using their non-dominant hand for the four different stimuli. Stroop Task results from these 30-s periods will not be taken into account so that participants can fill in the M-VAS scale and reset there focus on the Stroop Task. During each block, NIRS, HR, RR and SaO2 data will be assessed and averaged.

Control task:

In the control task subjects will have to watch a documentary during 60 min on the same computer screen as that used for the experimental trial. In order to avoid under- and over-arousal the subjects will have the opportunity to choose between several episodes (One Planet, Frozen Worlds, Jungles, Costal Seas, From Desserts to Grasslands, The High Seas, Fresh Water and Forests) of the Netflix documentary "Our Planet, 2019" as proposed by the research team. During the control task physiological and psychological measures will be assessed at the same time points as during the mental fatigue trial.

Time to exhaustion cycling test (TTE):

After completing the MF- or control task. Participants will be asked to take place on the (propositioned) cycle ergometer (Lode Excalibur Sport, Groningen, The Netherlands). After 2 minutes of passive sitting on the ergometer a 2-minute NIRS-baseline will be measured. When all baseline measures have been collected, participants will perform a 3-min warm-up at 40% of peak power output followed by a rectangular workload at a power output corresponding to their predetermined respiratory compensation point (±80% peak power output). Pedal frequency was freely chosen between 60 and 100 RPM and was recorded every minute. TTE was measured from the start of the rectangular workload until the pedal frequency was less than 60 RPM for more than 5 s despite standardized verbal encouragement provided by a research assistant blind to treatment allocation. This TTE task was chosen, based on a previous study of Marcora et al. (2009), who found that mental fatigue impairs physical performance. A researcher will sit behind the subject to ensure compliance with treatment. Subjects will be equipped with a heart rate monitor to continuously follow up heart rate (HR). Subjective psychological assessment will take place with a M-VAS-scale, the National Aeronautics and Space Administration Task Load Index (NASA-TLX), the success motivation and intrinsic motivation scales developed and validated by Matthews et al., Karolinska Sleepiness Scale (KSS) and visual analog scale for boredom (B-VAS).

ELIGIBILITY:
Inclusion Criteria:

* Healthy (No neurological or cardiovascular disorders)
* Male or female
* No medication
* Non-smoker • Between 18 and 35 years old
* Recreational athlete population; performance level 2 or 3 for men according to De Pauw et al. (2013)(De Pauw et al., 2013) and performance level 2 or 3 for woman according to Decroix et al. (2015)(Decroix et al., 2015)
* Non-acclimatized to altitude (at least 2 months)

Exclusion Criteria:

* Injuries
* Acclimated to altitude
* Use of medication
* Use of caffeine and heavy efforts 24 hours prior each trial
* Not eating a standardized meal, the morning of each trial

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2024-02-29 (Estimated); Study Completion 2024-02-29 (Estimated)

PRIMARY OUTCOMES:
Cerebral oxygenation | 2 hours
  Prefrontal cortex oxygenation = relative changes in oxy- and deoxy hemoglobin concentrations at the prefrontal cortex. During the whole frame, participants are equipped with a Near Infrared Spectroscopy device that measures cerebral oxygenation continuously at 10hz.
Mental Fatigue | 60 minutes
  Results of a visual analogue scale for mental fatigue (1 to 100) Higher score is more mentally fatigued
Time to exhaustion cycling | 1hour
  Cycling at a power output corresponding to the subject's respiratory compensation point until exhaustion

SECONDARY OUTCOMES:
Cognition | 7 minutes
  results of a computerized Go/NoGo task

OTHER OUTCOMES:
Hemoglobin concentration | 10 minutes
  Hemoglobin will be assessed through the analysys of 1 drop of arterial blood
Blood glucose concentration | 10 minutes
  Glucose will be assessed through the analysys of 1 drop of arterial blood
Blood Lactate concentration | 1 hour
  Blood lactate will be assessed through the analysys of 1 drop of arterial blood at the end of every 5-minute block of the time to exhaustion cycling task

CONTACTS AND LOCATIONS:
Locations (1):
- Human Physiology - MFYS, Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: Undecided